CLINICAL TRIAL: NCT02649322
Title: Randomized, Controlled Trial of Needleless Jet Injected (J-Tip) Lidocaine in Children Undergoing Regional Anesthesia Prior to Knee Arthroscopy.
Brief Title: Needleless Jet Injected (J-Tip) Lidocaine in Children Undergoing Regional Anesthesia Prior to Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Daryl Osbahr, Sports Medicine Orthopaedic physician, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14.099.08
Record Dates: First submitted 2015-12-13; First posted 2016-01-07 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Knee Injury
MeSH Terms: conditions — Knee Injuries | interventions — Syringes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants in Group A will receive 0.25 mL of 1% plain lidocaine delivered by the J-tip injector at the regional block site prior to introduction of the needle for the nerve block procedure.
  Interventions: Device: J-Tip
- Group B (Active Comparator): Participants in Group B will receive 2 mL of 1% plain lidocaine injected by syringe and 25 gauge needle at the regional block site prior to introduction of the needle for the nerve block procedure.
  Interventions: Device: Syringe and 25 gauge needle

INTERVENTIONS:
Device: J-Tip — After sterile preparation, the J-tip injector will be placed on the skin at the selected site of the regional block needle introduction. Firm pressure will be placed with the J-tip injector on the site for the chosen block, the safety ring slid down, the trigger pressed and the tip held firmly on the skin for three seconds. One quarter of a milliliter of one percent lidocaine will be injected with the characteristic "pop" and "hissing" sounds inherent to the J-tip injector.
  Arms: Group A
Device: Syringe and 25 gauge needle — The same initial timeout and sterile prep procedure will be followed for the use of local syringe and 25 gauge needle injection of 1% lidocaine ninety seconds prior to introduction of the regional block needle.
  Arms: Group B

SUMMARY:
Purpose of this study is to investigate the pain outcomes and satisfaction of pain relief for pediatric patients receiving needleless jet-injected (J-Tip) lidocaine prior to regional anesthesia with femoral and/or sciatic nerve block and general anesthesia for arthroscopic knee surgery compared to femoral nerve block and/or sciatic nerve block with needle injected lidocaine prior to regional and general anesthesia.

DETAILED DESCRIPTION:
The J-tip device has not been reported for use prior to regional block anesthesia prior to femoral or sciatic nerve blocks. The use of the J-tip device for lidocaine introduction prior to femoral or sciatic blocks at Arnold Palmer Medical Center has been up to the discretion of the anesthesiologist. It has been anecdotally reported at our institution to have equal or better pain relief for the regional nerve blocks as needle introduction of lidocaine.

This study seeks to evaluate the difference in pain from local anesthetic infiltration with J-tip needleless injection device compared to needle injection by use of Visual Analog Scales.

* To evaluate efficacy of femoral nerve block after J-tip device lidocaine injection post operatively by use of Visual Analog Scales.
* To assess patient and parent satisfaction with J-tip device use by satisfaction questionnaire.
* To assess changes in post operative pain medication amounts with J-tip device use.

ELIGIBILITY:
Inclusion Criteria:

Subjects between the ages of eleven and seventeen undergoing arthroscopic knee surgery.

* Able to independently complete the Visual Analog pain scales.
* Subjects who are neurologically intact at area of injection.
* English speaking.

Exclusion Criteria:

* Subjects with known allergies to lidocaine.
* Presence of developmental delay.
* Subjects with blood disorders affecting coagulation.
* Subjects on blood thinners.
* Subjects receiving chemotherapeutic agents.
* Those who use or receive analgesia prior to procedure, except for acetaminophen or Non-steroidal anti-inflammatory medications.
* Any other local sedation at the area of nerve block injection.
* Non-English Speaking
* Subjects with signs of skin infection or pathology at the injection site.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl C Osbahr, MD, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Lidocaine J-Tip: Participants in Group A will receive 0.25 mL of 1% plain lidocaine delivered by the J-tip injector at the regional block site prior to introduction of the needle for the nerve block procedure.
  J-Tip: After sterile preparation, the J-tip injector will be placed on the skin at the selected site of the regional block needle introduction. Firm pressure will be placed with the J-tip injector on the site for the chosen block, the safety ring slid down, the trigger pressed and the tip held firmly on the skin for three seconds. One quarter of a milliliter of one percent lidocaine will be injected with the characteristic "pop" and "hissing" sounds inherent to the J-tip injector.
- Group B Lidocaine Syringe: Participants in Group B will receive 2 mL of 1% plain lidocaine injected by syringe and 25 gauge needle at the regional block site prior to introduction of the needle for the nerve block procedure.
  Syringe and 25 gauge needle: The same initial timeout and sterile prep procedure will be followed for the use of local syringe and 25 gauge needle injection of 1% lidocaine ninety seconds prior to introduction of the regional block needle.
Period: Overall Study
Arm/Group | Group A Lidocaine J-Tip | Group B Lidocaine Syringe
Started | 58 | 57
Completed | 58 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Lidocaine J-Tip | Group B Lidocaine Syringe | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58 | 57 | 115
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15 [11 to 17] | 14 [11 to 17] | 15 [11 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 29 | 25 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 115
Participants [Count of Participants; unit: Participants] | 58 | 57 | 115

OUTCOME MEASURES:

1. Primary Outcome: Baseline Pain Assessment Before Knee Arthroscopy Via the Visual Analog Scale.
Description: Pain will be assessed via the Visual Analog Scale by the patient before administration of the nerve block. Patient will report on a scale of 0 to 10 what their perceived pain is. 0 is no pain with 10 being worst pain patient ever experienced.
Time Frame: During Baseline Assessment, Taking Approximately 20 Minutes, Before Nerve Block
Population: Comparison of the mean pain on visual analog scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A Lidocaine J-Tip | Group B Lidocaine Syringe
Number analyzed (Participants) | 58 | 57
score on a scale | .25 (1.243) | .43 (1.185)

2. Primary Outcome: Pain Assessment After Knee Arthroscopy Via the Visual Analog Scale
Description: Pain will be assess via the Visual Analog Scale by the patient after the knee arthroscopy though first post op office visit and average of one week. Patient will report on a scale of 0 to 10 what their perceived pain is. 0 is no pain with 10 being worst pain patient ever experienced.
Time Frame: During Follow-up Assessment at an Average of 1 Week Post Op
Population: Comparison of the mean pain on visual analog scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A Lidocaine J-Tip | Group B Lidocaine Syringe
Number analyzed (Participants) | 58 | 57
units on a scale | 1.54 (1.524) | 3.57 (2.133)

3. Secondary Outcome: Satisfaction Via a 0 to 10 Rating Scale at Follow up
Description: Patients will be asked to describe how satisfied they were with the knee arthroscopy via a 0 to 10 rating scale. Patient will report on a scale of 0 to 10 what their perceived satisfaction is. 0 is no satisfaction with 10 most satisfaction.
Time Frame: At the follow up appointment, an average of one week after the procedure.
Population: Comparison of the mean satisfaction on visual analog scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A Lidocaine J-Tip | Group B Lidocaine Syringe
Number analyzed (Participants) | 58 | 57
score on a scale | 2.384615385 (1.796149728) | 2.391304348 (2.623999904)

ADVERSE EVENTS:
Time Frame: 1 month post op
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 0/58 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT02649322/Prot_SAP_000.pdf